

## **NOTE TO FILE**

12-Jan-2018

Re: MLN1117-1501 SAP for ClinicalTrials.gov results submission

MLN1117-1501 was a 2-part (Phase 1/2) study. The Phase 1 portion of the study completed, but the Phase 2 portion of the study was cancelled though, due to decisions by the study team. Due to this early termination of the study, a statistical analysis plan was never drafted and analyses were not performed.